CLINICAL TRIAL: NCT02522104
Title: Evaluation of the Impact of Renal Function on the Pharmacokinetics of Hydroxyurea (SIKLOS ®) in Normal-renal Function, Hyperfiltrating and Renal Failure Sickle Cell Disease Patients (DARH)
Brief Title: Evaluation of the Impact of Renal Function on the Pharmacokinetics of SIKLOS ® (DARH)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Theravia (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SIK-FR 14-1
Record Dates: First submitted 2015-08-04; First posted 2015-08-13 (Estimated); Results first posted 2021-08-27 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-08

CONDITIONS: Sickle Cell Disease; Renal Function Disorder
Keywords: Pharmacokinetics of Hydroxyurea
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Hydroxyurea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Normal-renal function (Experimental): Normal-renal function: 90 ≤ GFR ≤ 130 mL/min/1.73m2 in women or 140 mL/min/1.73m2 in men
  Interventions: Drug: Siklos
- Glomerular hyperfiltration (Experimental): Glomerular renal hyperfiltration: GFR > 130 mL/min/1.73m2 in women and GFR > 140 mL/min/1.73m2 in men.
  Interventions: Drug: Siklos
- Moderate renal failure (Experimental): Moderate renal failure: 30 ≤ GFR ≤ 60 mL/min/1.73m2
  Interventions: Drug: Siklos

INTERVENTIONS:
Drug: Siklos
  Other Names: hydroxyurea

SUMMARY:
The use of hydroxyurea in sickle cell disease patients with glomerular hyperfiltration and renal failure requires a specific monitoring and dose adjustment in order to remain within the therapeutic interval while limiting the risk of toxicity or therapeutic failure. For this reason the investigators propose to compare the pharmacokinetic parameters of hydroxyurea in normal-renal function sickle cell patients to those of patients with glomerular hyperfiltration or moderate renal failure.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Male or female.
* Sickle cell disease (SS or S-β0thal) confirmed by haemoglobin electrophoresis and genotyping by deoxyribonucleic acid (DNA) analysis.
* Affiliation to a social security system.
* Having freely consented in writing after being informed of the objective, programme and potential risks incurred.

These criteria will apply to the 3 groups of sickle cell disease patients according to the renal function stage defined by the glomerular filtration rate (GFR) estimated by the formula of the Chronic Kidney Disease EPIdemiology (CKD EPI) collaboration without ethnic criterion during the last 6 months before inclusion:

* Normal-renal function: 90 ≤ GFR ≤ 130 mL/min/1.73m2 in women or 140 mL/min/1.73m2 in men.
* Moderate renal failure: 30 ≤ GFR ≤ 60 mL/min/1.73m2.
* Glomerular renal hyperfiltration: GFR > 130 mL/min/1.73m2 in women and GFR > 140 mL/min/1.73m2 in men.

  * Treated with hydroxyurea (Siklos®) with a stable dosage for at least one week ± 2 days before inclusion in the study and dose administered in the morning at 9:00 ± 15 minutes.

Exclusion Criteria:

* Refusal to consent.
* Patients that do not comply.
* Occurrence of vaso-occlusive crisis in the month prior to the inclusion in the study.
* Patients having had an exchange transfusion in the 15 days before inclusion in the study.
* Patients participating in another clinical trial or in the exclusion period of a previous clinical trial.
* Patients treated with a diuretic.
* Dialysis patient.
* Patients with an intercurrent disorder, especially inflammatory, that has not recovered for at least one month.
* Pregnant or breast-feeding women.
* Patients deprived of liberty or under legal protection.
* Patients who cannot understand the objective and the course of the study, incapable of giving their consent.
* In the event of severe hepatic failure.
* In the event of severe renal failure (creatinine clearance < 30 ml/min).
* Patients who show toxic signs of bone marrow suppression.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-09-03 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: BARTOLUCCI Pablo, MD, Principal Investigator — Centre de Référence des Syndromes Drépanocytaires Majeurs, Hôpital Henri-Mondor
Locations (1):
- Centre de Référence des Syndromes Drépanocytaires Majeurs, Hôpital Henri-Mondor, Créteil, France

RESULTS

PARTICIPANT FLOW:
Groups:
- Normal-renal Function: Patients with normal-renal function defined by 90 ≤ GFR ≤ 130 mL/min/1.73m2 in women or 140 mL/min/1.73m2 in men
- Glomerular Hyperfiltration: Patients with glomerular renal hyperfiltration defined by GFR > 130 mL/min/1.73m2 in women and GFR > 140 mL/min/1.73m2 in men
- Moderate Renal Failure: Patients with moderate renal failure defined by 30 ≤ GFR ≤ 60 mL/min/1.73m2
Period: Overall Study
Arm/Group | Normal-renal Function | Glomerular Hyperfiltration | Moderate Renal Failure
Started | 13 | 15 | 12
Completed | 10 | 12 | 5
Not Completed | 3 | 3 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal-renal Function | Glomerular Hyperfiltration | Moderate Renal Failure | Total
Number analyzed (Participants) | 10 | 12 | 5 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.2 (4.8) | 27.8 (7.6) | 50.0 (7.5) | 33.1 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 11 | 2 | 18
  Male | 5 | 1 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: Measure of Plasmatic Data: Maximum Concentration (Cmax)
Description: Compare the pharmacokinetic parameters of hydroxyurea in normal-renal function sickle cell patients to those of patients with glomerular hyperfiltration or moderate renal failure
Time Frame: 0 hour, 0.75 hour, 1.5 hours, 3 hours, 4 hours, 6 hours, 7.5 hours , 24 hours
Measure: Mean (Standard Deviation); unit: Micromolar
Arm/Group | Normal-renal Function | Glomerular Hyperfiltration | Moderate Renal Failure
Number analyzed (Participants) | 10 | 12 | 5
Micromolar | 271.8 (164.4) | 316.8 (73.9) | 260.2 (88.1)

2. Primary Outcome: Measure of Plasmatic Data: Minimum Concentration (Cmin)
Description: as for outcome 1
Time Frame: 0 hour, 0.75 hour, 1.5 hours, 3 hours, 4 hours, 6 hours, 7.5 hours , 24 hours
Measure: Mean (Standard Deviation); unit: Micromolar
Arm/Group | Normal-renal Function | Glomerular Hyperfiltration | Moderate Renal Failure
Number analyzed (Participants) | 10 | 12 | 5
Micromolar | 3.80 (2.38) | 4.2 (2.2) | 7.1 (4.4)

3. Primary Outcome: Measure of Plasmatic Data: Time to Obtain the Maximum Concentration (Tmax)
Description: as for outcome 1
Time Frame: 0 hour, 0.75 hour, 1.5 hours, 3 hours, 4 hours, 6 hours, 7.5 hours , 24 hours
Measure: Mean (Standard Deviation); unit: Hour
Arm/Group | Normal-renal Function | Glomerular Hyperfiltration | Moderate Renal Failure
Number analyzed (Participants) | 10 | 12 | 5
Hour | 0.9 (0.7) | 1.0 (0.9) | 1.0 (1.1)

4. Primary Outcome: Measure of Plasmatic Data: Area Under the Curve (AUC0-24)
Description: as for outcome 1
Time Frame: 0 hour, 0.75 hour, 1.5 hours, 3 hours, 4 hours, 6 hours, 7.5 hours , 24 hours
Measure: Mean (Standard Deviation); unit: Hour x Micromolar
Arm/Group | Normal-renal Function | Glomerular Hyperfiltration | Moderate Renal Failure
Number analyzed (Participants) | 10 | 12 | 5
Hour x Micromolar | 1144.0 (364.1) | 1384.3 (266.5) | 1580.6 (540.6)

5. Primary Outcome: Measure of Plasmatic Data: Elimination Half-life (T½)
Description: as for outcome 1
Time Frame: 0 hour, 0.75 hour, 1.5 hours, 3 hours, 4 hours, 6 hours, 7.5 hours , 24 hours
Measure: Mean (Standard Deviation); unit: Hour
Arm/Group | Normal-renal Function | Glomerular Hyperfiltration | Moderate Renal Failure
Number analyzed (Participants) | 10 | 12 | 5
Hour | 4.30 (0.57) | 4.75 (0.92) | 4.98 (0.90)

6. Primary Outcome: Measure of Plasmatic Data: Total Clearance (Cl Tot)
Description: as for outcome 1
Time Frame: 0 hour, 0.75 hour, 1.5 hours, 3 hours, 4 hours, 6 hours, 7.5 hours , 24 hours
Measure: Mean (Standard Deviation); unit: Liter/Hour
Arm/Group | Normal-renal Function | Glomerular Hyperfiltration | Moderate Renal Failure
Number analyzed (Participants) | 10 | 12 | 5
Liter/Hour | 10.1 (4.1) | 10.3 (1.9) | 6.4 (2.1)

7. Primary Outcome: Measure of Plasmatic Data: Distribution Volume
Description: as for outcome 1
Time Frame: 0 hour, 0.75 hour, 1.5 hours, 3 hours, 4 hours, 6 hours, 7.5 hours , 24 hours
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Normal-renal Function | Glomerular Hyperfiltration | Moderate Renal Failure
Number analyzed (Participants) | 10 | 12 | 5
Liter | 61.2 (20.3) | 70.3 (16.2) | 44.2 (11.4)

8. Primary Outcome: Measure of Urinary Data: Hydroxyurea Urinary Fractions
Description: as for outcome 1
Time Frame: From 0 to 4 hours, 4 to 7.5 hours and 7.5 to 24 hours
Measure: Mean (Standard Deviation); unit: Percentage urinary excretion
Arm/Group | Normal-renal Function | Glomerular Hyperfiltration | Moderate Renal Failure
Number analyzed (Participants) | 10 | 12 | 5
Percentage urinary excretion | 35.8 (10.2) | 44.3 (9.6) | 20.2 (7.3)

9. Primary Outcome: Measure of Urinary Data: Renal Clearance (Cl Renal).
Description: as for outcome 1
Time Frame: From 0 to 4 hours, 4 to 7.5 hours and 7.5 to 24 hours
Measure: Mean (Standard Deviation); unit: Liter/Hour
Arm/Group | Normal-renal Function | Glomerular Hyperfiltration | Moderate Renal Failure
Number analyzed (Participants) | 10 | 12 | 5
Liter/Hour | 3.9 (1.6) | 4.7 (1.3) | 1.3 (0.7)

ADVERSE EVENTS:
Time Frame: From the signature of the informed consent form by the patient until 7 days after the end of the follow-up for the study. Duration of participation for each patients : 9 to 40 days depending on the concomitant treatments.
Arm/Group | Normal-renal Function | Glomerular Hyperfiltration | Moderate Renal Failure
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/12 | 0/5
Serious Adverse Events (participants affected / at risk) | 1/10 | 0/12 | 1/5
Other Adverse Events (participants affected / at risk) | 2/10 | 0/12 | 0/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Normal-renal Function (N=10) | Glomerular Hyperfiltration (N=12) | Moderate Renal Failure (N=5)
Aplastic anemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Hypotension (Cardiac disorders) | 1 | 0 | 0
Vaso-occlusive crisis (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Normal-renal Function (N=10) | Glomerular Hyperfiltration (N=12) | Moderate Renal Failure (N=5)
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fever (General disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No